CLINICAL TRIAL: NCT01273064
Title: A Placebo-Controlled, Multicenter, Double-Blind, Randomized Trial of Pegylated Interferon Plus Ribavirin With or Without CTS-1027 in HCV Null-Responders
Brief Title: Standard of Care (SOC) With or Without CTS-1027 in Hepatitis C (HCV) Null-Responders
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Risk-benefit ratio
Sponsor: Conatus Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTS-1027-05
Record Dates: First submitted 2010-12-21; First posted 2011-01-10 (Estimated); Results first posted 2012-05-30 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Hepatitis C
Keywords: HCV; Null Responders
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- CTS-1027 60 mg + ribavirin + peglyated interferon (Experimental): Standard of Care (ribavirin plus pegylated interferon) plus CTS-1027, 60 mg (supplied in a blinded kit containing two bottles of 30 mg tablets). One tablet from each of the CTS bottles is taken twice daily, for a total daily dose of 120 mg.
  Interventions: Drug: CTS-1027; Drug: pegylated interferon; Drug: Ribavirin
- CTS-1027 30 mg + ribavirin + pegylated interferon (Experimental): Standard of Care (ribavirin plus pegylated interferon) plus CTS-1027 30 mg, supplied in a blinded kit containing one bottle of 30 mg tablets, and one bottle of placebo tablets (in order to maintain blind). One tablet from each of the bottles is taken twice daily, for a total daily dose of 60 mg of CTS-1027.
  Interventions: Drug: CTS-1027; Drug: pegylated interferon; Drug: Ribavirin; Drug: Placebo
- CTS-1027 15 mg + ribavirin + pegylated interferon (Experimental): Standard of Care (ribavirin plus pegylated interferon) plus CTS-1027 15 mg (supplied in a blinded kit containing one bottle each of of 5 mg and 10 mg tablets). One tablet from each of the CTS bottles is taken twice daily, for a total daily dose of 30 mg.
  Interventions: Drug: CTS-1027; Drug: pegylated interferon; Drug: Ribavirin
- placebo + ribavirin + pegylated interferon (Active Comparator): Standard of Care (ribavirin plus pegylated interferon) plus placebo (supplied in a blinded kit containing two bottles of placebo tablets). One tablet is taken from each of the placebo bottles twice daily, for a total daily dose of 4 tablets.
  Interventions: Drug: pegylated interferon; Drug: Ribavirin; Drug: Placebo

INTERVENTIONS:
Drug: CTS-1027 — Supplied in 30mg, 10mg, or 5mg tablets (depending on dose arm) taken twice daily for up to 48 weeks.
  Arms: CTS-1027 15 mg + ribavirin + pegylated interferon; CTS-1027 30 mg + ribavirin + pegylated interferon; CTS-1027 60 mg + ribavirin + peglyated interferon
Drug: pegylated interferon — 180 micrograms in 0.5 ml of solution subcutaneously (SQ), delivered in single use syringes administered once per week, for up to 48 weeks.
  Other Names: Pegasys
Drug: Ribavirin — 200 mg capsules of ribavirn taken in two divided daily doses totaling 1000 mg (5 capsules) for patients weighing 75 kg or less, or 1200 mg (6 capsules) for patients weighing more than 75 kg
  Other Names: Copegus
Drug: Placebo — Tablets identical in appearance to CTS-1027 containing inactive ingredients.
  Placebo arm patients: Two tablets taken twice daily, for a total daily dose of four tablets.
  30 mg CTS-1027 patients: One tablet taken twice daily, for a total daily dose of two tablets. One bottle of placebo is added to the 30mg kits in order to maintain the study blind (all patients recieve two-bottle kits of CTS-1027 and/or placebo).
  Arms: CTS-1027 30 mg + ribavirin + pegylated interferon; placebo + ribavirin + pegylated interferon

SUMMARY:
Placebo controlled, double-blind, multicenter study utilizing standard of care (SOC) treatment (ribavirin plus pegylated interferon) in combination with CTS-1027 in genotype 1 chronic Hepatitis C (HCV) patients who were null-responders to previous SOC therapy(ies).

Null-responders are defined as patients who failed to achieve a greater than 2 log drop in HCV-RNA (Hepatitis C Ribonucleic acid, also known as "viral load") levels after 12 weeks of treatment (know as an "early virologic response", or EVR) during previous SOC therapy.

If, during previous SOC treatment, a patient had a less than 2 log decline in HCV-RNA at Week 12 but greater than 2 log decline in HCV-RNA at any time from Week 12 to Week 24, that patient is not a null-responder, and is excluded from study participation. If, during previous SOC treatment, a Week 12 HCV-RNA was not obtained, the post Week 12 response must have been < 2 log decline (and still HCV-RNA positive) in order for the patient to be defined as a null-responder.

Patients will be screened and have up to 4 weeks to qualify for study entry. During this screening period, clinical and laboratory tests will be performed. At Week 0/Day 1, patients will undergo centralized, stratified (based on ethnicity), randomization to one of four treatment arms: SOC + one of three doses of CTS-1027 or SOC + placebo. Study treatment will last 24, 48, or 60 weeks, based on each patient's response to study treatment. SOC + placebo patients who do not show a virologic response after 12 weeks of therapy will be rolled onto SOC + 15mg CTS-1027, while maintaining the study blind.

DETAILED DESCRIPTION:
Placebo controlled, double-blind, multicenter study utilizing Standard of Care (SOC) in combination with CTS-1027 in genotype 1 chronic hepatitis C (HCV) patients who were null-responders to previous SOC therapy(ies).

Null-responders are defined as patients who failed to achieve a greater than 2 log drop in HCV-RNA levels after 12 weeks of treatment (know as an early virologic response or EVR) during previous SOC therapy.

If, during previous SOC treatment, a patient had < 2 log decline in HCV-RNA at Week 12 but > 2 log decline in HCV-RNA at any time from Week 12 to Week 24, that patient is not a null-responder and is excluded from study participation. If, during previous SOC treatment, a Week 12 HCV-RNA was not obtained, the post Week 12 response must have been < 2 log decline (and still HCV-RNA positive) in order for the patient to be defined as a null-responder.

Patients will be screened and have up to 4 weeks to qualify for study entry. During this screening period, clinical and laboratory tests will be performed. At Week 0/Day 1, patients will undergo centralized, stratified (based on ethnicity), randomization to one of four treatment arms: SOC + one of three doses of CTS-1027 or SOC + placebo. Study treatment will last 24, 48, or 60 weeks, based on each patient's response to study treatment.

The Principal Investigators, other site personnel, and patients will be blinded to the HCV-RNA results for the first 12 weeks of therapy.

At Week 12, the study treatment blind will be broken by the study's Interactive Web Randomization System (IWRS). However, the Principal Investigators, other investigative site personnel, patients, and Sponsor will remain blinded to treatment allocation until Week 24 (see below). The patients on the SOC + placebo arm will continue treatment as follows:

* Patients on SOC + placebo who do not achieve at least a 2 log decline in their HCV-RNA at Week 12 will be automatically rolled-over into the SOC + 15 mg CTS-1027 twice a day (BID) arm. The treatment duration for these patients will be 60 weeks (i.e., 12 weeks on SOC + placebo, followed by 48 weeks on SOC + 15 mg BID).
* Those patients on SOC + placebo who achieve ≥ 2 log decline at Week 12 will continue on SOC therapy until Week 48.

Patients in the SOC + CTS-1027 arms will continue with the same treatment regimen for the initial 24 weeks regardless of HCV-RNA changes.

At Week 24, the study blind will be formally broken. Patients will continue the study as follows:

* Patients in the SOC + CTS-1027 arms who achieve ≥ 2 log HCV-RNA decline by Week 24 will continue with the same treatment regimen they were assigned during the Double-Blind Phase for an additional 24 weeks.
* Patients in the SOC + CTS-1027 15 mg BID and the SOC + CTS-1027 30 mg BID arms who achieve a <2 log HCV-RNA decline by Week 24 will escalate to the next higher dose of CTS-1027 for an additional 24 weeks.
* Patients in the SOC + CTS-1027 60 mg BID arm who do not achieve at least a 2 log HCV-RNA decline by Week 24 will be discontinued from the study.

All patients will be seen 4 and 12 weeks (Follow-Up Period) after the end of treatment. If a patient's HCV-RNA is undetectable at the end of treatment, he/she will be seen for an additional follow-up visit 24 weeks after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients of minimum adult legal age (according to local laws for signing the informed consent document), able to provide written informed consent, and understand and comply with the requirements of the study
2. HCV genotype 1 infected null responders to prior therapy comprised of pegylated interferon and ribavirin (standard of care, SOC) defined as:

   * Failure to achieve an early virologic response (< 2 log decline in HCV-RNA by Week 12), or
   * If Week 12 HCV-RNA was not obtained, post Week 12 HCV-RNA response was < 2 log decline
3. Screening HCV-RNA viral load of > 5.0 log (i.e., >100,000 IU/mL)
4. alpha-fetoprotein (AFP) less than or equal to 100 ng/mL
5. Hemoglobin greater than or equal to 12 g/dL for women and greater than or equal to 13 g/dL for men, hemoglobin A1c less than or equal to 7.5 %, platelet count greater than or equal to 90 x 10^9/L, and white blood cell count greater than or equal to 1.5 x 10^9/L
6. Thyroid Stimulating Hormone (TSH) within normal limits
7. In the opinion of the Principal Investigator, the patient met the 80%/80%/80% rule during the previous pegylated interferon and ribavirin therapy (i.e., received at least 80% of the pegylated interferon and ribavirin doses, at least 80% of the dose size, for at least 80% of the treatment duration)
8. Willingness to utilize two reliable forms of contraception (for both males and females of childbearing potential) from screening to at least six months after the completion of the study.

Exclusion Criteria:

1. < 2 log decline in HCV-RNA at Week 12 but > 2 log decline at any time from Week 12 to Week 24 during prior therapy with pegylated interferon and ribavirin (prior standard of care therapy)
2. Decompensated or severe liver disease defined by one or more of the following criteria:

   * Prothrombin time 4 seconds > control or INR (international normalized ratio) > 1.2
   * Total bilirubin ≥ 1.5 mg/dL or direct bilirubin ≥ 1 mg/dL
   * Serum albumin below normal limits
   * aspartate aminotransferase (AST) or alanine aminotransferase (ALT)> 5 x upper limit of normal (ULN) at screening
   * Presence of ascites
3. Hepatic encephalopathy
4. Hepatocellular carcinoma (HCC) or suspicion of HCC clinically or on ultrasound (or other imaging techniques)
5. Clinically significant ocular findings such as retinopathy, cotton wool spots, optic nerve disorder, retinal hemorrhage, or other abnormality
6. Known history or presence of human immunodeficiency virus (HIV) infection
7. Co-infection with hepatitis B virus (HBV)
8. If female: pregnant, lactating, or positive serum or urine pregnancy test
9. Male partners of women who are currently pregnant
10. Renal impairment (creatinine > 1.2 x ULN), serum creatinine clearance < 50 mL/min, or hepatorenal syndrome with ascites
11. Hospitalization for liver disease within 60 days of screening
12. History of alcohol abuse (> 50 g per day) within the past year
13. History of severe psychiatric disease, especially depression, characterized by:

    * Suicide attempt
    * Hospitalization for psychiatric disease
    * Period of disability as a result of psychiatric disease
14. Prior exposure to CTS-1027
15. Patients who qualify as a null-responder based on treatment(s) other than pegylated interferon and ribavirin
16. History or presence of clinically concerning cardiac arrhythmias or prolongation of pre-dose corrected Q-T interval (QTc) of > 450 milliseconds
17. History of or current autoimmune disease
18. Diagnosis of or symptoms suggestive of fibromyalgia
19. Currently on liver transplantation waiting list or recipient of any organ transplant
20. Other concomitant disease or condition likely to significantly decrease life expectancy (e.g., moderate to severe congestive heart failure) or any malignancy other than curatively treated skin cancer (basal cell or squamous cell carcinomas), unless adequately treated or in complete remission for five or more years
21. Exposure to any other investigational treatment for any aspect of disease associated with HCV during the past 6 months
22. Exposure to any investigational drug or device within 30 days of dosing, or scheduled receipt of another investigational drug or device during the course of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Castelloe, MD, Study Chair — Conatus Pharmaceuticals Inc.
Locations (45):
- United States (45):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Southern California Liver Centers, Coronado, California
  - Scripps Clinic, La Jolla, California
  - Loma Linda University MC, Loma Linda, California
  - Huntington Medical Research Institute, Pasadena, California
  - Medical Associates Research Group, San Diego, California
  - UCSD, San Diego, California
  - University of Colorado Denver, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - Atlanta Medical Center, Inc., Atlanta, Georgia
  - Liver Center of Atlanta, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Loyola University, Maywood, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - St. Louis University, St Louis, Missouri
  - Concorde Medical Group, New York, New York
  - New York University, New York, New York
  - Weill Medical College of Cornell, New York, New York
  - Columbia Presbyterian Medical Center, New York, New York
  - Einstein College of Medicine (Jacobi Medical Center), The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Duke University Medical Center, Durham, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Baylor All Saints Medical Center, Fort Worth, Texas
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - Research Specialists of Texas, Houston, Texas
  - St. Luke's Episcopal Hospital, Houston, Texas
  - University of Texas HSC at Houston, Houston, Texas
  - VAMC Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Metropolitan Research Group Washington DC, Fairfax, Virginia
  - Liver Institute of Virginia, Newport News, Virginia
  - Virginia Commonwealth University (VCU), Richmond, Virginia
  - Benaroya Research Institute at Virginia Mason, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- CTS-1027 60 mg + Ribavirin + Peglyated Interferon: Standard of Care (ribavirin plus pegylated interferon) plus CTS-1027,60 mg (supplied in 30 mg tablets) taken twice daily, for a total daily dose of 120 mg
- CTS-1027 30 mg + Ribavirin + Pegylated Interferon: Standard of Care (ribavirin plus pegylated interferon) plus CTS-1027 30 mg (supplied in 30 mg tablets) taken twice daily for a total daily dose of 60 mg.
- CTS-1027 15 mg + Ribavirin + Pegylated Interferon: Standard of Care (ribavirin plus pegylated interferon) plus CTS-1027 15 mg (supplied in 5 mg and 10 mg tablets) taken twice daily, for a total daily dose of 30 mg
- Placebo + Ribavirin + Pegylated Interferon: Standard of Care (ribavirin plus pegylated interferon) plus placebo (2 tablets identical in appearance to CTS-1027) taken twice daily, for a total daily dose of 4 tablets
- Placebo + CTS-1027 15mg + Ribavirin + Pegylated Interferon: Standard of Care (ribavirin plus pegylated interferon) plus placebo (2 tablets identical in appearance to CTS-1027) taken twice daily, for a total daily dose of 4 tablets for the first 12 weeks. Crossover to Standard of Care (ribavirin plus pegylated interferon) plus CTS-1027 15mg (supplied in 5 mg and 10 mg tablets) taken twice daily, for a total daily dose of 30 mg starting at Week 12
Period: Overall Study
Arm/Group | CTS-1027 60 mg + Ribavirin + Peglyated Interferon | CTS-1027 30 mg + Ribavirin + Pegylated Interferon | CTS-1027 15 mg + Ribavirin + Pegylated Interferon | Placebo + Ribavirin + Pegylated Interferon | Placebo + CTS-1027 15mg + Ribavirin + Pegylated Interferon
Started | 23 | 30 | 31 | 20 | 10 (Began study on the placebo arm, and crossed over to CTS-1027 15 mg at Wk 12 due to lack of response)
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 23 | 30 | 31 | 20 | 10
Not completed — Adverse Event | 5 | 1 | 3 | 2 | 1
Not completed — Withdrawal by Subject | 4 | 2 | 2 | 2 | 0
Not completed — Study Termination | 13 | 27 | 26 | 16 | 8
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CTS-1027 60 mg + Ribavirin + Peglyated Interferon | CTS-1027 30 mg + Ribavirin + Pegylated Interferon | CTS-1027 15 mg + Ribavirin + Pegylated Interferon | Placebo + Ribavirin + Pegylated Interferon | Placebo + CTS-1027 15mg + Ribavirin + Pegylated Interferon | Total
Number analyzed (Participants) | 23 | 30 | 31 | 20 | 10 | 114
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 29 | 28 | 20 | 8 | 108
  >=65 years | 0 | 1 | 3 | 0 | 2 | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 53.1 (7.0) | 55.1 (6.0) | 50.5 (11.3) | 52.8 (7.1) | 57.7 (5.9) | 53.2 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 12 | 6 | 3 | 41
  Male | 13 | 20 | 19 | 14 | 7 | 73
Region of Enrollment [Number; unit: participants]
  United States | 23 | 30 | 31 | 20 | 10 | 114

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virologic Response
Description: Percent of patients that achieve a sustained virologic response (SVR) at Week 72 defined as HCV-RNA (Hepatitis C virus ribonucleic acid, also known as 'viral load') level below the quantification limit (BQL) at Week 72.
Time Frame: Baseline and 24 weeks after the end of treatment (Week 72)
Population: Due to the premature discontinuation of this study and termination of the entire CTS-1027 program, an efficacy analysis was not conducted. No patients completed the study.
Measure: Number; unit: Percent of participants
Arm/Group | CTS-1027 60 mg + Ribavirin + Peglyated Interferon | CTS-1027 30 mg + Ribavirin + Pegylated Interferon | CTS-1027 15 mg + Ribavirin + Pegylated Interferon | Placebo + Ribavirin + Pegylated Interferon | Placebo + CTS-1027 15mg + Ribavirin + Pegylated Interferon
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Greater Than 2 Log Decline in HCV-RNA at Study Weeks 12, 24 and 48
Description: Percent of patients experiencing a drop in Hepatitis C virus ribonucleic acid (HCV-RNA, also known as "viral load") levels in the blood equal to, or greater than, 2 log from before treatment (baseline) through 12, 24, and 48 weeks of treatment.
Time Frame: Baseline, and Study Weeks 12, 24, and 48
Population: as for outcome 1
Measure: Number; unit: Percent of participants
Arm/Group | CTS-1027 60 mg + Ribavirin + Peglyated Interferon | CTS-1027 30 mg + Ribavirin + Pegylated Interferon | CTS-1027 15 mg + Ribavirin + Pegylated Interferon | Placebo + Ribavirin + Pegylated Interferon | Placebo + CTS-1027 15mg + Ribavirin + Pegylated Interferon
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 of dosing through 4 to 12 weeks after treatment discontinuation.
Description: Adverse events listed are those reported by at least 5% of the patients, and deemed potentially related (possibly, probably, or definitely) to study any of the medications by the Investigator. All serious adverse events are reported regardless of causality.
Arm/Group | CTS-1027 60 mg + Ribavirin + Peglyated Interferon | CTS-1027 30 mg + Ribavirin + Pegylated Interferon | CTS-1027 15 mg + Ribavirin + Pegylated Interferon | Placebo + Ribavirin + Pegylated Interferon | Placebo + CTS-1027 15mg + Ribavirin + Pegylated Interferon
Serious Adverse Events (participants affected / at risk) | 2/23 | 0/30 | 0/31 | 1/20 | 1/10
Other Adverse Events (participants affected / at risk) | 23/23 | 28/30 | 26/31 | 19/20 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CTS-1027 60 mg + Ribavirin + Peglyated Interferon (N=23) | CTS-1027 30 mg + Ribavirin + Pegylated Interferon (N=30) | CTS-1027 15 mg + Ribavirin + Pegylated Interferon (N=31) | Placebo + Ribavirin + Pegylated Interferon (N=20) | Placebo + CTS-1027 15mg + Ribavirin + Pegylated Interferon (N=10)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enteritis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholestatic liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CTS-1027 60 mg + Ribavirin + Peglyated Interferon (N=23) | CTS-1027 30 mg + Ribavirin + Pegylated Interferon (N=30) | CTS-1027 15 mg + Ribavirin + Pegylated Interferon (N=31) | Placebo + Ribavirin + Pegylated Interferon (N=20) | Placebo + CTS-1027 15mg + Ribavirin + Pegylated Interferon (N=10)
Anemia (Blood and lymphatic system disorders) | 4 (4) | 5 (5) | 2 (2) | 1 (1) | 3 (4)
Neutopenia (Blood and lymphatic system disorders) | 2 (2) | 4 (4) | 2 (2) | 2 (2) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 3 (5) | 4 (6) | 2 (2) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (8) | 9 (11) | 7 (8) | 6 (9) | 4 (5)
Asthenia (General disorders) | 3 (3) | 2 (2) | 0 (0) | 4 (5) | 0 (0)
Chills (General disorders) | 4 (5) | 5 (5) | 2 (2) | 2 (2) | 2 (2)
Fatigue (General disorders) | 15 (17) | 16 (19) | 12 (14) | 8 (8) | 6 (7)
Influenza like illness (General disorders) | 1 (1) | 4 (5) | 4 (4) | 4 (4) | 0 (0)
Injection site erythema (General disorders) | 1 (2) | 2 (2) | 1 (1) | 2 (2) | 1 (3)
Injection site reaction (General disorders) | 2 (2) | 3 (4) | 0 (0) | 1 (1) | 0 (0)
Irritability (General disorders) | 4 (5) | 6 (7) | 4 (4) | 2 (2) | 1 (3)
Pain (General disorders) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 4 (5) | 3 (5) | 3 (4) | 0 (0)
Decreased appetite (General disorders) | 6 (8) | 6 (6) | 3 (3) | 2 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (15) | 13 (14) | 5 (6) | 1 (2) | 4 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4) | 1 (1) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 7 (9) | 5 (6) | 2 (2) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 3 (4) | 2 (2) | 4 (4) | 6 (6) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 9 (9) | 9 (9) | 12 (16) | 10 (12) | 5 (5)
Anxiety (Psychiatric disorders) | 1 (2) | 3 (4) | 2 (2) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 4 (5) | 4 (4) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (6) | 8 (12) | 5 (6) | 3 (3) | 4 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 1 (1) | 2 (2) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3) | 5 (5) | 1 (1) | 3 (3)
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hyperhirosis (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (8) | 5 (6) | 3 (3) | 1 (1) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (3) | 8 (8) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
This study was terminated early after 3 reports of hyperbilirubinemia occurred(2 on 60mg bid and 1 on 30mg bid of CTS 1027). Two incidents were reported as part of an SAE. The risk/benefit ratio did not warrant further continuation of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less